CLINICAL TRIAL: NCT06919809
Title: Efficacy and Safety of X A-DERM™ Microsurfaced Acellular Dermal Matrix (mADM) for Enhancing Wound Healing Following Mohs Micrographic Surgery (MMS)
Brief Title: Effectiveness and Safety of X A-DERM™ Microsurfaced Acellular Dermal Matrix for Wound Healing After MOHS Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGuire Institute (Industry)
Collaborators: CellTherX (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTX2025-01
Record Dates: First submitted 2025-03-28; First posted 2025-04-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Wound Healing After MMS Surgery; BCC - Basal Cell Carcinoma; SCC - Squamous Cell Carcinoma; Melanoma In Situ
Keywords: MMS; BCC; SCC; MIS; Melanoma In Situ; Wound Healing; Scar Quality; Wound Management; Wound Cosmetics
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Recipient of the X A-DERM™ mADM (Experimental): The participants will receive the X A-DERM™ mADM following MMS for removal of BCC, SCC, or MIS lesions in the face, head, or upper extremities. After complete excision of the tumor and removal of all cancerous tissue, reconstruction immediately follows with placement of the mADM into the defect. Subjects will receive the standard of care for post-op and at-home wound care and will be recalled for a total of 5 in-office visits to evaluate wound healing.
  Interventions: Device: A microsurfaced ADM (acellular dermal matrix)

INTERVENTIONS:
Device: A microsurfaced ADM (acellular dermal matrix) — X A-DERM™ ADM has been resurfaced (Microsurfaced) instead of currently utilized smooth surface reconstructive grafts. Microsurfacing of regenerative tissue grafts increases the surface area at the graft-to-host interface and results in quicker absorption of blood into the graft, greater cellular infiltration, improved seal and wound bed preparedness.
  Other Names: X A-DERM™ ADM

SUMMARY:
The goal of this single-arm clinical trial is to learn about the effectiveness and safety of the X A-DERM™ mADM in promoting wound healing and improving scar formation after MMS surgery for removing BCC, SCC, or MIS lesions on the face, head, and upper limbs. The main questions it aims to answer are how well this intervention works and what is the safety profile.

The primary hypothesis is that the use of X A-DERM™ will result improved wound healing and scar formation after 60 days post-procedure.

Participants will undergo MMS surgery to remove BCC, SCC, or MIS lesions, and then will receive the X A-DERM™ mADM graft at the surgical site. Participants will return to the office four additional times for the clinician to collect data on their wound healing. This will involve taking pictures of the wound, conducting clinical assessments (CROs), and documenting the patient's reported outcomes (PROs).

DETAILED DESCRIPTION:
The objective of this trial is to evaluate the efficacy and safety of X A-DERM™ mADM for enhancing wound healing and improving scar formation following MMS for removal of BCC, SCC, or MIS lesions in the face, head, upper and lower extremities, and trunk in adults 18 to 85 years of age who are scheduled to undergo elective MMS. After complete excision of the tumor and removal of all cancerous tissue, reconstruction immediately follows with placement of the mADM into the defect. Subjects will receive the standard of care for post-op and at-home wound care and will be recalled for a total of 5 in-office visits to evaluate wound healing. This is a single-arm, open-label, prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all the following criteria to be entered into the study:

1. Between 18 and 85 years of age, inclusive
2. Subject in good health, or with stable treated medical condition, as determined by the investigator.
3. Scheduled to undergo elective Mohs surgery to remove a single biopsy-proven basal cell carcinoma (BCC), squamous cell carcinoma (SCC), or melanoma in situ (MIS) lesion on the head, face, or upper extremity that is amenable to Mohs surgery.
4. Tumor location and size meets the following criteria for immediate MMS:

   * Largest total surface area of ≤16cm2 and smallest total surface area per PI discretion.
   * Depth with majority of tumor excision at least to subcutaneous tissue.
   * Adequate dermal contract with graft.
5. Willing and able to complete and comply with procedures, protocol requirements, and instructions, including self-performed wound care and completion of all required visits.
6. Able to speak, read, write, and understand the language of the informed consent form (ICF) and study questionnaires.
7. Willingness and ability to understand the risks, benefits, and alternatives to participation, and give informed consent.

   -

Exclusion Criteria: Subjects who meet the above inclusion criteria will be eligible for the study, unless they present with any of the following:

1. History of wound abnormalities or any other findings that would impede participation in the trial, as per PI discretion.
2. Post-operative defects superficial and deemed not appropriate for second intention healing, as determined by the investigator.
3. Pregnant, lactating/breast feeding, or planning a pregnancy. A negative urine pregnancy test will be required at screening for female subjects of childbearing potential; a woman will be considered to be of childbearing potential unless she has had a tubal ligation, total hysterectomy, bilateral oophorectomy, or is postmenopausal (without a menstrual period for at least one year).

   -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of X A-DERM™ mADM on clinician- and patient-based assessments and objective measurements of wound healing and scar quality. | Visit 1(Day 0), Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 30), and Visit 5 (Day 60).
  This will be done by capturing digital photographs. Digital photographs of the wound bed site will be acquired pre- and post-placement of the mADM perioperatively and at follow-up visits.
To evaluate the effectiveness of X A-DERM™ mADM on clinician- and patient-based assessments and objective measurements of wound healing and scar quality. | Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 30), and Visit 5 (Day 60).
  This will be done by requesting patients and clinicians to complete POSAS assessments, the Patient and Observer Scar Assessment Scale. The POSAS contains two assessments. The first assessment captures patients' views on scar pain, itchiness, if the scar color is different, if the scar is more stiff, is the thickness of the scar different, and is the scar irregular by ranking their answer from a scale of 1-10. 1 being "no, no complaints" and 10 being "yes, worst imaginable". The second assessment is the clinician's portion. It involves objective scoring based on standardized criteria for characteristics such as vascularity, pigmentation, thickness, relief, pliability, and surface area using a scale from 1-10 1 being "Normal skin" and 10 being "worst scar imaginable".

SECONDARY OUTCOMES:
To evaluate the effectiveness of X A-DERM™ mADM on objective metrics of wound healing based on physical measurements as well as subjective assessments on wound management, pain, functional outcomes, quality of life, and cosmetic appearance | Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 30), and Visit 5 (Day 60).
  This will be done by completing clinician reported outcomes. The first clinician reported outcome tool used is the Visual Analog Scale (VAS) for scar appearance. It is completed by making a mark across the line corresponding to the clinician observation between the statements at each of the extremes. The associated "lines" encapsulate a spectrum of scar appearance with "excellent" on one end and "poor" on the opposite.
To evaluate the effectiveness of X A-DERM™ mADM on objective metrics of wound healing based on physical measurements as well as subjective assessments on wound management, pain, functional outcomes, quality of life, and cosmetic appearance | Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 30), and Visit 5 (Day 60).
  This will be done by completing clinician reported outcomes. The second clinician reported outcome tool used is the Manchester Scar Satisfaction Scale (MSSS). It is completed by the clinician evaluating the patient's scar by checking the box of the corresponding characteristic that best matches their assessment for 5 parameters. The first parameter is color (compared to surrounding skin), and the options are perfect, slight mismatch, obvious mismatch, and gross mismatch. The second matte or shiny, and those are the two options. The third is contour, the options being flush with surrounding area, slightly proud (indented), hypertrophic, and keloid. The fourth is distortion with options of none, mild, moderate, and severe. The last parameter is texture with options of normal, just palpable, firm, and hard.
To evaluate the effectiveness of X A-DERM™ mADM on objective metrics of wound healing based on physical measurements as well as subjective assessments on wound management, pain, functional outcomes, quality of life, and cosmetic appearance | Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 30), and Visit 5 (Day 60).
  This will be done by completing patient reported outcomes. The first patient reported outcome tool used is the Visual Analog Scale (VAS) for pain intensity, itching intensity, and cosmetic appearance. It is completed by the patient making a mark across the line corresponding to their observation between the statements at each of the extremes. The associated "lines" encapsulate a spectrum of pain intensity ("no pain" and "worst pain imaginable"), itching intensity ("no itch" and "worst itch imaginable"), and cosmetic appearance ("worst scar" and "best scar").
To evaluate the effectiveness of X A-DERM™ mADM on objective metrics of wound healing based on physical measurements as well as subjective assessments on wound management, pain, functional outcomes, quality of life, and cosmetic appearance | Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 30), and Visit 5 (Day 60).
  This will be done by completing patient reported outcomes. The second patient reported outcome tool used is the ease of wound care numerical rating scale (NRS). The patient reports on a scale from 0 to 10, where 0 represents "Very Easy" and 10 represents "Impossible," please rate how easy it was for them to care for the wound by themself?
To evaluate the effectiveness of X A-DERM™ mADM on objective metrics of wound healing based on physical measurements as well as subjective assessments on wound management, pain, functional outcomes, quality of life, and cosmetic appearance | Visit 2 (Day 7), Visit 3 (Day 14), Visit 4 (Day 30), and Visit 5 (Day 60).
  This will be done by completing patient reported outcomes. The third patient reported outcome tool used is the Skindex-16 questionnaire. The patient will for each of the following questions, make a mark in the box corresponding to your feelings about each of the statements. The scale is "never bothered" to "always bothered" on a 0-6 numerical rank and the various conditions are as follows: itching, burning or stinging, hurting, your skin condition being irritated, the persistence/reoccurrence of your skin condition, worry about your skin condition, the appearance, frustration, embarrassment, being annoyed about your skin condition, feeling depressed about your skin condition, the effects of your skin condition on your desire to be with people, your skin condition making it hard to show affection, the effects of your skin condition on your daily activities, and your skin condition making it hard to work or do what you enjoy.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Drake, Study Director — CellTherX; Aaron Farberg, MD, Principal Investigator — Bare Dermatology
Locations (1):
- Bare Dermatology, Rockwall, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data. Results will be published in peer-reviewed journals, with aggregate data only.

REFERENCES:
- [Background] Commander SJ, Chamata E, Cox J, Dickey RM, Lee EI. Update on Postsurgical Scar Management. Semin Plast Surg. 2016 Aug;30(3):122-8. doi: 10.1055/s-0036-1584824. PMID 27478420
- [Background] Broughton G 2nd, Janis JE, Attinger CE. The basic science of wound healing. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):12S-34S. doi: 10.1097/01.prs.0000225430.42531.c2. PMID 16799372
- [Background] Rubin DB. Multiple imputation for nonresponse in surveys. Hoboken, N.J. ;: Wiley-Interscience; 2004: xxix, 287 p.
- [Background] Schafer JL. Analysis of Incomplete Multivariate Data: CRC Press; 1997.
- [Background] Allison PD. Missing Data: SAGE Publications; 2001.
- [Background] National Research Council (US) Panel on Handling Missing Data in Clinical Trials. The Prevention and Treatment of Missing Data in Clinical Trials. Washington (DC): National Academies Press (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK209904/ PMID 24983040
- [Background] West BT, Welch KB, Gałecki AT, Gillespie BW. Linear mixed models : a practical guide using statistical software. Boca Raton: CRC Press, Taylor & Francis Group; 2015: xxv, 414 pages.
- [Background] Goldstein H. Multilevel statistical models. Chichester, West Sussex: Wiley; 2011: xxi, 358 p.
- [Background] Gilthorpe MS, Dahly DL, Tu YK, Kubzansky LD, Goodman E. Challenges in modelling the random structure correctly in growth mixture models and the impact this has on model mixtures. J Dev Orig Health Dis. 2014 Jun;5(3):197-205. doi: 10.1017/S2040174414000130. PMID 24901659
- [Background] EMA. Guideline On Adjustment for Baseline Covariates in Clinical Trials (EMA/CHMP/295050/2013). In: Use EMACfMPfH, ed.: European Medicines Agency Amsterdam, 2013.
- [Background] Cheng J, Edwards LJ, Maldonado-Molina MM, Komro KA, Muller KE. Real longitudinal data analysis for real people: building a good enough mixed model. Stat Med. 2010 Feb 20;29(4):504-20. doi: 10.1002/sim.3775. PMID 20013937
- [Background] Maxwell SE, Kelley K, Rausch JR. Sample size planning for statistical power and accuracy in parameter estimation. Annu Rev Psychol. 2008;59:537-63. doi: 10.1146/annurev.psych.59.103006.093735. PMID 17937603
- [Background] Phillips A, Abellan-Andres J, Soren A, Bretz F, Fletcher C, France L, Garrett A, Harris R, Kjaer M, Keene O, Morgan D, O'Kelly M, Roger J. Estimands: discussion points from the PSI estimands and sensitivity expert group. Pharm Stat. 2017 Jan;16(1):6-11. doi: 10.1002/pst.1745. Epub 2016 Mar 21. PMID 26997517
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Background] FDA. Guidance for Industry - Non-Inferiority Clinical Trials to Establish Effectiveness. No. Food and Drug Administration, 2016. (U.S. Department of Health and Human Services publication
- [Background] EMA. Points to Consider on Switching between Superiority and Non-Inferiority (CPMP/EWP/482/99). In: Products EMACfPM, ed.: European Medicines Agency London, 2000
- [Background] EMA. Guideline on the Choice of the Non-Inferiority Margin (EMEA/CPMP/EWP/2158/99). In: Use EMACfMPfH, ed.: European Medicines Agency London, 2006.
- [Background] Badersten A, Nilveus R, Egelberg J. Effect of nonsurgical periodontal therapy. I. Moderately advanced periodontitis. J Clin Periodontol. 1981 Feb;8(1):57-72. doi: 10.1111/j.1600-051x.1981.tb02024.x. PMID 6972954
- [Background] PASS. Power Analysis and Sample Size Software. In. Kaysville, Utah, USA: NCSS, LLC, 2023.
- [Background] Gergely LH, Gaspar K, Brodszky V, Kinyo A, Szegedi A, Remenyik E, Kiss NF, Bato A, Pentek M, Gulacsi L, Sardy M, Banvolgyi A, Wikonkal N, Rencz F. Validity of EQ-5D-5L, Skindex-16, DLQI and DLQI-R in patients with hidradenitis suppurativa. J Eur Acad Dermatol Venereol. 2020 Nov;34(11):2584-2592. doi: 10.1111/jdv.16642. Epub 2020 Jul 2. PMID 32618022
- [Background] Chren MM, Lasek RJ, Sahay AP, Sands LP. Measurement properties of Skindex-16: a brief quality-of-life measure for patients with skin diseases. J Cutan Med Surg. 2001 Mar-Apr;5(2):105-10. doi: 10.1007/BF02737863. Epub 2001 Mar 21. PMID 11443481
- [Background] Chren MM. The Skindex instruments to measure the effects of skin disease on quality of life. Dermatol Clin. 2012 Apr;30(2):231-6, xiii. doi: 10.1016/j.det.2011.11.003. Epub 2011 Dec 20. PMID 22284137
- [Background] Chren MM, Lasek RJ, Quinn LM, Covinsky KE. Convergent and discriminant validity of a generic and a disease-specific instrument to measure quality of life in patients with skin disease. J Invest Dermatol. 1997 Jan;108(1):103-7. doi: 10.1111/1523-1747.ep12285650. PMID 8980297
- [Background] Chren MM, Lasek RJ, Flocke SA, Zyzanski SJ. Improved discriminative and evaluative capability of a refined version of Skindex, a quality-of-life instrument for patients with skin diseases. Arch Dermatol. 1997 Nov;133(11):1433-40. PMID 9371029
- [Background] Reich A, Heisig M, Phan NQ, Taneda K, Takamori K, Takeuchi S, Furue M, Blome C, Augustin M, Stander S, Szepietowski JC. Visual analogue scale: evaluation of the instrument for the assessment of pruritus. Acta Derm Venereol. 2012 Sep;92(5):497-501. doi: 10.2340/00015555-1265. PMID 22102095
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Quinn JV, Drzewiecki AE, Stiell IG, Elmslie TJ. Appearance scales to measure cosmetic outcomes of healed lacerations. Am J Emerg Med. 1995 Mar;13(2):229-31. doi: 10.1016/0735-6757(95)90100-0. PMID 7893315
- [Background] Quinn JV, Drzewiecki A, Li MM, Stiell IG, Sutcliffe T, Elmslie TJ, Wood WE. A randomized, controlled trial comparing a tissue adhesive with suturing in the repair of pediatric facial lacerations. Ann Emerg Med. 1993 Jul;22(7):1130-5. doi: 10.1016/s0196-0644(05)80977-1. PMID 8517562
- [Background] Panchapakesan V, Klassen AF, Cano SJ, Scott AM, Pusic AL. Development and psychometric evaluation of the FACE-Q Aging Appraisal Scale and Patient-Perceived Age Visual Analog Scale. Aesthet Surg J. 2013 Nov 1;33(8):1099-109. doi: 10.1177/1090820X13510170. Epub 2013 Nov 15. PMID 24243890
- [Background] Beausang E, Floyd H, Dunn KW, Orton CI, Ferguson MW. A new quantitative scale for clinical scar assessment. Plast Reconstr Surg. 1998 Nov;102(6):1954-61. doi: 10.1097/00006534-199811000-00022. PMID 9810991
- [Background] Masters M, McMahon M, Svens B. Reliability testing of a new scar assessment tool, Matching Assessment of Scars and Photographs (MAPS). J Burn Care Rehabil. 2005 May-Jun;26(3):273-84. PMID 15879752
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Schneider CA, Rasband WS, Eliceiri KW. NIH Image to ImageJ: 25 years of image analysis. Nat Methods. 2012 Jul;9(7):671-5. doi: 10.1038/nmeth.2089. PMID 22930834
- [Background] Schindelin J, Arganda-Carreras I, Frise E, Kaynig V, Longair M, Pietzsch T, Preibisch S, Rueden C, Saalfeld S, Schmid B, Tinevez JY, White DJ, Hartenstein V, Eliceiri K, Tomancak P, Cardona A. Fiji: an open-source platform for biological-image analysis. Nat Methods. 2012 Jun 28;9(7):676-82. doi: 10.1038/nmeth.2019. PMID 22743772
- [Background] Bien P, De Anda C, Prokocimer P. Comparison of digital planimetry and ruler technique to measure ABSSSI lesion sizes in the ESTABLISH-1 study. Surg Infect (Larchmt). 2014 Apr;15(2):105-10. doi: 10.1089/sur.2013.070. Epub 2014 Jan 22. PMID 24450727
- [Background] Chang AC, Dearman B, Greenwood JE. A comparison of wound area measurement techniques: visitrak versus photography. Eplasty. 2011 Apr 18;11:e18. PMID 21559060
- [Background] Treuillet S, Albouy B, Lucas Y. Three-dimensional assessment of skin wounds using a standard digital camera. IEEE Trans Med Imaging. 2009 May;28(5):752-62. doi: 10.1109/TMI.2008.2012025. Epub 2009 Jan 13. PMID 19150787
- [Background] Foltynski P, Ladyzynski P, Ciechanowska A, Migalska-Musial K, Judzewicz G, Sabalinska S. Wound Area Measurement with Digital Planimetry: Improved Accuracy and Precision with Calibration Based on 2 Rulers. PLoS One. 2015 Aug 7;10(8):e0134622. doi: 10.1371/journal.pone.0134622. eCollection 2015. PMID 26252747
- [Background] Foltynski P, Ladyzynski P. Digital Planimetry With a New Adaptive Calibration Procedure Results in Accurate and Precise Wound Area Measurement at Curved Surfaces. J Diabetes Sci Technol. 2022 Jan;16(1):128-136. doi: 10.1177/1932296820959346. Epub 2020 Oct 1. PMID 33000645
- [Background] Foltynski P. Ways to increase precision and accuracy of wound area measurement using smart devices: Advanced app Planimator. PLoS One. 2018 Mar 5;13(3):e0192485. doi: 10.1371/journal.pone.0192485. eCollection 2018. PMID 29505569
- [Background] Goldman RJ, Salcido R. More than one way to measure a wound: an overview of tools and techniques. Adv Skin Wound Care. 2002 Sep-Oct;15(5):236-43. doi: 10.1097/00129334-200209000-00011. PMID 12368715
- [Background] Gilman T. Wound outcomes: the utility of surface measures. Int J Low Extrem Wounds. 2004 Sep;3(3):125-32. doi: 10.1177/1534734604264419. PMID 15866803
- [Background] Gronbeck C, Beltrami EJ, Jain N, Hargis G, Sloan B, Cook BL, Grant-Kels JM, Feng H. Surface anatomy in dermatology: Part II-Impact on perioperative management, procedural technique, and cosmesis. J Am Acad Dermatol. 2024 Aug;91(2):223-240. doi: 10.1016/j.jaad.2023.07.002. Epub 2023 Jul 8. PMID 37429437
- [Background] Beltrami EJ, Gronbeck C, Jain N, Hargis G, Feng H, Grant-Kels JM, Sloan B. Surface anatomy in dermatology: Part I-Clinical importance, diagnostic utility, and impact on medical management. J Am Acad Dermatol. 2024 Aug;91(2):207-220. doi: 10.1016/j.jaad.2023.07.001. Epub 2023 Jul 8. PMID 37429436
- [Background] Strobl KH, Hirzinger G. More accurate pinhole camera calibration with imperfect planar target. In: 2011 IEEE International Conference on Computer Vision Workshops (ICCV Workshops), 2011:1068-1075.
- [Background] Rogers LC, Bevilacqua NJ, Armstrong DG, Andros G. Digital planimetry results in more accurate wound measurements: a comparison to standard ruler measurements. J Diabetes Sci Technol. 2010 Jul 1;4(4):799-802. doi: 10.1177/193229681000400405. PMID 20663440
- [Background] Moore K. Using wound area measurement to predict and monitor response to treatment of chronic wounds. J Wound Care. 2005 May;14(5):229-32. doi: 10.12968/jowc.2005.14.5.26771. PMID 15909440
- [Background] Bloemen MC, Boekema BK, Vlig M, van Zuijlen PP, Middelkoop E. Digital image analysis versus clinical assessment of wound epithelialization: a validation study. Burns. 2012 Jun;38(4):501-5. doi: 10.1016/j.burns.2012.02.003. Epub 2012 Feb 29. PMID 22381563
- [Background] Jorgensen LB, Sorensen JA, Jemec GB, Yderstraede KB. Methods to assess area and volume of wounds - a systematic review. Int Wound J. 2016 Aug;13(4):540-53. doi: 10.1111/iwj.12472. Epub 2015 Aug 6. PMID 26250714
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Durani P, McGrouther DA, Ferguson MW. Current scales for assessing human scarring: a review. J Plast Reconstr Aesthet Surg. 2009 Jun;62(6):713-20. doi: 10.1016/j.bjps.2009.01.080. Epub 2009 Mar 20. PMID 19303834
- [Background] Legemate CM, Middelkoop E, Carriere ME, van Zuijlen PPM, van Baar ME, van der Vlies CH; Hycon Study group. The minimal important change (MIC) and minimal clinically important difference (MCID) of the patient and observer scar assessment scale (POSAS) 2.0. Burns. 2024 Nov;50(8):2070-2076. doi: 10.1016/j.burns.2024.05.022. Epub 2024 Jun 6. PMID 38902132
- [Background] Durani P, McGrouther DA, Ferguson MW. The Patient Scar Assessment Questionnaire: a reliable and valid patient-reported outcomes measure for linear scars. Plast Reconstr Surg. 2009 May;123(5):1481-1489. doi: 10.1097/PRS.0b013e3181a205de. PMID 19407619
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Wainwright D, Madden M, Luterman A, Hunt J, Monafo W, Heimbach D, Kagan R, Sittig K, Dimick A, Herndon D. Clinical evaluation of an acellular allograft dermal matrix in full-thickness burns. J Burn Care Rehabil. 1996 Mar-Apr;17(2):124-36. doi: 10.1097/00004630-199603000-00006. PMID 8675502
- [Background] Alam M, Ibrahim O, Nodzenski M, Strasswimmer JM, Jiang SI, Cohen JL, Albano BJ, Batra P, Behshad R, Benedetto AV, Chan CS, Chilukuri S, Crocker C, Crystal HW, Dhir A, Faulconer VA, Goldberg LH, Goodman C, Greenbaum SS, Hale EK, Hanke CW, Hruza GJ, Jacobson L, Jones J, Kimyai-Asadi A, Kouba D, Lahti J, Macias K, Miller SJ, Monk E, Nguyen TH, Oganesyan G, Pennie M, Pontius K, Posten W, Reichel JL, Rohrer TE, Rooney JA, Tran HT, Poon E, Bolotin D, Dubina M, Pace N, Kim N, Disphanurat W, Kathawalla U, Kakar R, West DP, Veledar E, Yoo S. Adverse events associated with mohs micrographic surgery: multicenter prospective cohort study of 20,821 cases at 23 centers. JAMA Dermatol. 2013 Dec;149(12):1378-85. doi: 10.1001/jamadermatol.2013.6255. PMID 24080866
- [Background] Sclafani AP, Sclafani JA, Sclafani AM. Successes, revisions, and postoperative complications in 446 Mohs defect repairs. Facial Plast Surg. 2012 Jun;28(3):358-66. doi: 10.1055/s-0032-1312691. Epub 2012 Jun 21. PMID 22723239
- [Background] Cook JL, Perone JB. A prospective evaluation of the incidence of complications associated with Mohs micrographic surgery. Arch Dermatol. 2003 Feb;139(2):143-52. doi: 10.1001/archderm.139.2.143. PMID 12588220
- [Background] Mordick TG, Hamilton R, Dzubow LM. Delayed reconstruction following Mohs' chemosurgery for skin cancers of the head and neck. Am J Surg. 1990 Oct;160(4):447-9. doi: 10.1016/s0002-9610(05)80563-x. PMID 2221253
- [Background] WOOD WB Jr. Phagocytosis, with particular reference to encapsulated bacteria. Bacteriol Rev. 1960 Mar;24(1):41-9. doi: 10.1128/br.24.1.41-49.1960. No abstract available. PMID 13845837
- [Background] Teh BT. Why do skin grafts fail? Plast Reconstr Surg. 1979 Mar;63(3):323-32. doi: 10.1097/00006534-197903000-00005. PMID 368835
- [Background] Burleson R, Eiseman B. Mechanisms of antibacterial effect of biologic dressings. Ann Surg. 1973 Feb;177(2):181-6. doi: 10.1097/00000658-197302000-00010. No abstract available. PMID 4572783
- [Background] Marinelli L. ea. Histologic Evaluation of Wound-Bed Preparedness Following Microsurfaced Skin Grafts for the Treatment of Deep Burn Wounds: Results from a Randomized Controlled Trial. In: Professionals TSoFH, ed. Association of Military Surgeons of the United States (AMSUS) Annual Meeting. National Harbor, MD, 2023
- [Background] Tolkachjov SN, Brodland DG, Coldiron BM, Fazio MJ, Hruza GJ, Roenigk RK, Rogers HW, Zitelli JA, Winchester DS, Harmon CB. Understanding Mohs Micrographic Surgery: A Review and Practical Guide for the Nondermatologist. Mayo Clin Proc. 2017 Aug;92(8):1261-1271. doi: 10.1016/j.mayocp.2017.04.009. PMID 28778259
- [Background] Ferrari B, Reggiani C, Francomano M, Bellini P, Ferrari F, Giacomelli L, Mannocci A, Magnoni C. Clinical Factors Influencing the Outcomes of an Acellular Dermal Matrix for Skin Cancer Treatment: A Retrospective Study. Adv Skin Wound Care. 2020 Jul;33(7):367-374. doi: 10.1097/01.ASW.0000666900.03111.c3. PMID 32544116
- [Background] Lewis RE, Towery EA, Bhat SG, Ward AJ, Heidel RE, Bielak KM, Simpson HE, McLoughlin JM, Lewis JM. Human Acellular Dermal Matrix Is a Viable Alternative to Autologous Skin Graft in Patients with Cutaneous Malignancy. Am Surg. 2019 Sep 1;85(9):1056-1060. PMID 31638524
- [Background] Ravitskiy L, Brodland DG, Zitelli JA. Cost analysis: Mohs micrographic surgery. Dermatol Surg. 2012 Apr;38(4):585-94. doi: 10.1111/j.1524-4725.2012.02341.x. Epub 2012 Mar 22. PMID 22443180
- [Background] Tognetti L, Pianigiani E, Ierardi F, Lorenzini G, Casella D, Liso FG, De Pascalis A, Cinotti E, Rubegni P. The use of human acellular dermal matrices in advanced wound healing and surgical procedures: State of the art. Dermatol Ther. 2021 Jul;34(4):e14987. doi: 10.1111/dth.14987. Epub 2021 May 24. PMID 33993627
- [Background] Melman L, Jenkins ED, Hamilton NA, Bender LC, Brodt MD, Deeken CR, Greco SC, Frisella MM, Matthews BD. Early biocompatibility of crosslinked and non-crosslinked biologic meshes in a porcine model of ventral hernia repair. Hernia. 2011 Apr;15(2):157-64. doi: 10.1007/s10029-010-0770-0. Epub 2011 Jan 8. PMID 21222009
- [Background] Clark RA, Ghosh K, Tonnesen MG. Tissue engineering for cutaneous wounds. J Invest Dermatol. 2007 May;127(5):1018-29. doi: 10.1038/sj.jid.5700715. PMID 17435787
- [Background] Cho SK, Mattke S, Gordon H, Sheridan M, Ennis W. Development of a Model to Predict Healing of Chronic Wounds Within 12 Weeks. Adv Wound Care (New Rochelle). 2020 Sep;9(9):516-524. doi: 10.1089/wound.2019.1091. Epub 2020 Jan 24. PMID 32941121
- [Background] Cammarata E, Esposto E, Airoldi C, Giorgione R, Boggio P, Savoia P. Mohs micrographic technique in high-risk basal cell carcinoma: a 3D prediction of safety margins. J Wound Care. 2024 Aug 1;33(Sup8a):cxciv-cxcviii. doi: 10.12968/jowc.2020.0322. PMID 39163154
- [Background] Castillo J, Fathi R, McIlwee B, Williams K. Before and After Mohs Surgery: What to Expect for Patients. In: (ACMS) ACoMS, ed.: American College of Mohs Surgery Foundation's Mohs Surgeons Leading the Future (MSLF) Program., 2017:https://online.flippingbook.com/view/502707499/.
- [Background] Zurcher S, Martignoni Z, Hunger RE, Benzaquen M, Seyed Jafari SM. Mohs Micrographic Surgery for Cutaneous Squamous Cell Carcinoma. Cancers (Basel). 2024 Jun 28;16(13):2394. doi: 10.3390/cancers16132394. PMID 39001454
- [Background] Hong SN, Le Van D, Ngan GP, et al. MOHS MICROGRAPHIC SURGERY FOR BASAL CELL CARCINOMA: A REVIEW OF TREATMENT RESULTS. Tạp chí Da liễu học Việt Nam 2023.
- [Background] Wood LD, Ammirati CT. An overview of Mohs micrographic surgery for the treatment of basal cell carcinoma. Dermatol Clin. 2011 Apr;29(2):153-60, vii. doi: 10.1016/j.det.2011.02.005. PMID 21421141
- [Background] van Loo E, Mosterd K, Krekels GA, Roozeboom MH, Ostertag JU, Dirksen CD, Steijlen PM, Neumann HA, Nelemans PJ, Kelleners-Smeets NW. Surgical excision versus Mohs' micrographic surgery for basal cell carcinoma of the face: A randomised clinical trial with 10 year follow-up. Eur J Cancer. 2014 Nov;50(17):3011-20. doi: 10.1016/j.ejca.2014.08.018. Epub 2014 Sep 25. PMID 25262378
- [Background] Rowe DE, Carroll RJ, Day CL Jr. Long-term recurrence rates in previously untreated (primary) basal cell carcinoma: implications for patient follow-up. J Dermatol Surg Oncol. 1989 Mar;15(3):315-28. doi: 10.1111/j.1524-4725.1989.tb03166.x. PMID 2646336
- [Background] Snow SN, Larson PO, Lucarelli MJ, Lemke BN, Madjar DD. Sebaceous carcinoma of the eyelids treated by mohs micrographic surgery: report of nine cases with review of the literature. Dermatol Surg. 2002 Jul;28(7):623-31. doi: 10.1046/j.1524-4725.2002.01306.x. PMID 12135523
- [Background] American Academy of Dermatology; American College of Mohs Surgery; American Society for Dermatologic Surgery Association; American Society for Mohs Surgery; Ad Hoc Task Force; Connolly SM, Baker DR, Coldiron BM, Fazio MJ, Storrs PA, Vidimos AT, Zalla MJ, Brewer JD, Begolka WS, Berger TG, Bigby M, Bolognia JL, Brodland DG, Collins S, Cronin TA Jr, Dahl MV, Grant-Kels JM, Hanke CW, Hruza GJ, James WD, Lober CW, McBurney EI, Norton SA, Roenigk RK, Wheeland RG, Wisco OJ. AAD/ACMS/ASDSA/ASMS 2012 appropriate use criteria for Mohs micrographic surgery: a report of the American Academy of Dermatology, American College of Mohs Surgery, American Society for Dermatologic Surgery Association, and the American Society for Mohs Surgery. Dermatol Surg. 2012 Oct;38(10):1582-603. doi: 10.1111/j.1524-4725.2012.02574.x. Epub 2012 Sep 7. PMID 22958088
- [Background] Rogers HW, Weinstock MA, Harris AR, Hinckley MR, Feldman SR, Fleischer AB, Coldiron BM. Incidence estimate of nonmelanoma skin cancer in the United States, 2006. Arch Dermatol. 2010 Mar;146(3):283-7. doi: 10.1001/archdermatol.2010.19. PMID 20231499
- [Background] Miller SJ, Alam M, Andersen J, Berg D, Bichakjian CK, Bowen G, Cheney RT, Glass LF, Grekin RC, Kessinger A, Lee NY, Liegeois N, Lydiatt DD, Michalski J, Morrison WH, Nehal KS, Nelson KC, Nghiem P, Olencki T, Perlis CS, Rosenberg EW, Shaha AR, Urist MM, Wang LC, Zic JA. Basal cell and squamous cell skin cancers. J Natl Compr Canc Netw. 2010 Aug;8(8):836-64. doi: 10.6004/jnccn.2010.0062. No abstract available. PMID 20870631
- [Background] Miller SJ, Alam M, Andersen J, Berg D, Bichakjian CK, Bowen G, Cheney RT, Glass F, Grekin RC, Grichnik JM, Kessinger A, Lee NY, Lessin S, Lydiatt DD, Margolis LW, Michalski J, Nehal KS, Nghiem P, Oseroff AR, Rosenberg EW, Shaha AR, Siegle RJ, Urist MM; National Comprehensive Cancer Network. Basal cell and squamous cell skin cancers. J Natl Compr Canc Netw. 2007 May;5(5):506-29. doi: 10.6004/jnccn.2007.0045. No abstract available. PMID 17509254
- [Background] Lane JE, Kent DE. Surgical margins in the treatment of nonmelanoma skin cancer and mohs micrographic surgery. Curr Surg. 2005 Sep-Oct;62(5):518-26. doi: 10.1016/j.cursur.2005.01.003. PMID 16125611
- [Background] Gamret AC, Roberts JE, Srivastava D, Nijhawan RI. Mohs Micrographic Surgery: A Brief Overview. Semin Plast Surg. 2024 Nov 4;38(4):264-267. doi: 10.1055/s-0044-1791563. eCollection 2024 Nov. PMID 39697403
- [Background] Donaldson MR, Coldiron BM. Scars after second intention healing. Facial Plast Surg. 2012 Oct;28(5):497-503. doi: 10.1055/s-0032-1325643. Epub 2012 Oct 1. PMID 23027216
- See also: Related Info — https://celltherx.com/